CLINICAL TRIAL: NCT04038060
Title: Evaluation of Stepped PrEP (Pre-exposure Prophylaxis) Adherence Support for Young South African Women Using a SMART Design
Brief Title: The PrEP (Pre-exposure Prophylaxis) SMART Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Wits Reproductive Health and HIV Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Connie Celum, Prof of Medicine & Global Health, Adjunct Prof of Epidemiology, University of Washington
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00006439; R01MH114544 (NIH)
Record Dates: First submitted 2019-06-19; First posted 2019-07-30 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: HIV/AIDS
Keywords: pre-exposure prophylaxis; young women; HIV infections/prevention; SMART design
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Intervention Model Description: Sequential multiple assignment randomized trial (SMART)
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- WhatsApp Group (Experimental): Participants will be assigned to participate in a WhatsApp Group
  Interventions: Behavioral: WhatsApp Group
- 2-way SMS (Experimental): Participants will be assigned to receive weekly 2-way SMS initiated by the study team
  Interventions: Behavioral: 2-way SMS
- 2-way SMS and monthly counseling sessions (Experimental): Participants will be assigned to receive weekly 2-way SMS initiated by the study team and monthly counseling sessions
  Interventions: Behavioral: 2-way SMS; Behavioral: Monthly counseling sessions
- 2-way SMS and drug level feedback (Experimental): Participants will be assigned to receive weekly 2-way SMS initiated by the study team and drug level feedback
  Interventions: Behavioral: 2-way SMS; Behavioral: Drug level feedback
- WhatsApp Group and monthly counseling sessions (Experimental): Participants will be assigned to participate in a WhatsApp Group and monthly counseling sessions
  Interventions: Behavioral: WhatsApp Group; Behavioral: Monthly counseling sessions
- WhatsApp Group and drug level feedback (Experimental): Participants will be assigned to participate in a WhatsApp Group and drug level feedback
  Interventions: Behavioral: WhatsApp Group; Behavioral: Drug level feedback

INTERVENTIONS:
Behavioral: WhatsApp Group — Participants will receive peer adherence support through WhatsApp groups
  Arms: WhatsApp Group; WhatsApp Group and drug level feedback; WhatsApp Group and monthly counseling sessions
Behavioral: 2-way SMS — Participants will receive healthcare worker adherence support through 2-way SMS
  Arms: 2-way SMS; 2-way SMS and drug level feedback; 2-way SMS and monthly counseling sessions
Behavioral: Drug level feedback — Participants will receive adherence counseling based on tenofovir drug levels
  Arms: 2-way SMS and drug level feedback; WhatsApp Group and drug level feedback
Behavioral: Monthly counseling sessions — Participants will receive monthly counseling on a variety of issues that may be impacting their PrEP adherence
  Arms: 2-way SMS and monthly counseling sessions; WhatsApp Group and monthly counseling sessions

SUMMARY:
The PrEP SMART study is testing a stepped model of scalable adherence support strategies in South African young women who initiate PrEP using a SMART (sequential multiple assignment randomized trial) design.

DETAILED DESCRIPTION:
Women enrolled in the study will be randomized to standard of care adherence support (brief counseling) and either WhatsApp groups or weekly two-way SMS messages. Two months after PrEP initiation, tenofovir drug levels will be measured to determine if participants have achieved high adherence based on their initial randomization. Women with high adherence (i.e., TFV-DP >/=500 fmol/punch from dried blood spots [DBS]) will continue with the adherence support to which they were initially randomized. Participants with low adherence (i.e., TFV-DP <500 fmol/punch from DBS) will continue initial randomization (WhatsApp or two-way SMS) plus be randomized to more one of two more intensive adherence support interventions - continued monthly visits with adherence and problem-focused counseling at months 3-8 or quarterly visits between months 3-9 with feedback about adherence based on drug levels at months 3 and 6.

ELIGIBILITY:
Inclusion Criteria:

* Female at birth
* Age 18-25 years
* Per participant report, sexually active, defined as having vaginal or anal intercourse at least once in the month prior to screening
* Literate in one or more of the study languages
* Willing and able to provide informed consent
* Able and willing to provide adequate locator information
* Regular access to a mobile phone with SMS and WhatsApp capacity
* Agrees not to participate in other research studies involving drugs or medical devices for the duration of study participation

Exclusion Criteria:

* Planning to relocate in the next 12 months
* Has a job or other obligations that would require long absences from the area (> 4 weeks at a time) for 12 months
* A reactive or positive HIV test at Enrollment
* Any reported PrEP use within the last 6 months
* Concomitant participation in a clinical trial using investigational agents, including placebo-controlled clinical trials using such agents
* Prior participation in the active arm, or current participation in any arm, of an HIV vaccine trial
* Positive pregnancy test

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
PrEP Adherence | 9 months
  Evaluation of the proportion of young women who adhere well to PrEP in each of the intervention arms.

SECONDARY OUTCOMES:
PrEP persistence | 12 months
  Assessment of the proportion of young women who achieve high adherence.
Correlates of PrEP adherence | 12 months
  Assessment of the correlates of PrEP adherence, after adjusting for study arm.
PrEP discontinuation | 12 months
  Assessment of the timing of PrEP discontinuation in young women who discontinue PrEP.
PrEP decision making | 12 months
  Qualitative exploration of the factors that influence women's decisions to adhere to PrEP.
Intervention satisfaction | 12 months
  Qualitative exploration of women's satisfaction with their assigned intervention(s).

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, MD, MPH, Principal Investigator — University of Washington; Sinead Delany-Moretlwe, MBChB, PhD, Principal Investigator — Wits Reproductive Health and HIV Institute
Locations (1):
- Wits Reproductive Health and HIV Institute, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data from the PrEP SMART Study will be available at the end of the project by contacting the Principal Investigators.

REFERENCES:
- [Derived] Velloza J, Poovan N, Meisner A, Ndlovu N, Ndimande-Khoza N, Grabow C, Zwane P, Mbele S, Molefe M, Donnell D, Baeten JM, Hosek S, Celum C, Delany-Moretlwe S. Adaptive HIV pre-exposure prophylaxis adherence interventions for young women in Johannesburg, South Africa: a sequential multiple-assignment randomised trial. Lancet HIV. 2025 Feb;12(2):e105-e117. doi: 10.1016/S2352-3018(24)00268-6. Epub 2024 Dec 13. PMID 39681126
- [Derived] Velloza J, Poovan N, Ndlovu N, Khoza N, Morton JF, Omony J, Mkwanazi E, Grabow C, Donnell D, Munthali R, Baeten JM, Hosek S, Celum C, Delany-Moretlwe S. Adaptive HIV pre-exposure prophylaxis adherence interventions for young South African women: Study protocol for a sequential multiple assignment randomized trial. PLoS One. 2022 Apr 13;17(4):e0266665. doi: 10.1371/journal.pone.0266665. eCollection 2022. PMID 35417485